CLINICAL TRIAL: NCT01362582
Title: Open-label Randomized Multicentre Phase IIIb Trial Comparing Parenteral Substitution Versus Best Supportive Nutritional Care in Patients With Pancreatic Cancer Receiving 2nd Line Chemotherapy
Brief Title: Comparing Parenteral Nutrition vs Best Supportive Nutritional Care in Patients With Pancreatic Cancer
Acronym: PANUSCO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2008-11-03-1018; 60516908 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2010-11-25; First posted 2011-05-30 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; progression under chemotherapy; parenteral nutrition; pancreatic adenocarcinoma; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy, Nutritional Care (No Intervention): 5-Fluorouracil (5-FU) 2000mg/m2 IV (24-hour)/folinic acid (FA) 200mg/m2 IV (30 min) will be administered weekly over four weeks with additional oxaliplatin 85 mg/m2 IV (2-hour) on days 8 and 22. Therapy will be interrupted between days 23 to 42. The next cycle will be started on day 43.
  Subjects in the control group receive Best Supportive Nutritional Care. BSNC is defined as nutritional consultation and recommendation by experienced ecotrophologists.
- PN, Chemotherapy, Nutritional Care (Experimental): 5-Fluorouracil (5-FU) 2000mg/m2 IV (24-hour)/folinic acid (FA) 200mg/m2 IV (30 min) will be administered weekly over four weeks with additional oxaliplatin 85 mg/m2 IV (2-hour) on days 8 and 22. Therapy will be interrupted between days 23 to 42. The next cycle will be started on day 43.
  Patients receive also Best Supportive Nutritional Care defined as nutritional consultation and recommendation by experienced ecotrophologists.
  Intervention: Supportive Parenteral Nutrition
  Interventions: Drug: SMOF Kabiven

INTERVENTIONS:
Drug: SMOF Kabiven — SMOFKabiven® will be given over night with a content of 1100 kcal in 986 ml.
  Arms: PN, Chemotherapy, Nutritional Care

SUMMARY:
A randomised multicentre clinical phase IIIb trial for patients suffering from pancreatic adenocarcinoma receiving defined second or higher line chemotherapy and additionally parenteral nutrition (study arm A) or best supportive nutritional care (study arm B).

DETAILED DESCRIPTION:
Pancreatic cancer is an extremely aggressive malignancy characterized by extensive invasion, early metastasis, and marked cachexia. Subjects are afflicted with a variety of disconcerting symptoms, including profound cachexia and deterioration in performance status, even when their tumour burden is low. Therefore, one of the most important therapeutic targets is the improvement of quality of life. Supplementation with parenteral nutrition improves Quality of Life in subjects with advanced cancer cachexia. The European Society of Parenteral and Enteral Nutrition recommend PN only for malnourished subjects but does not reflect situation in cancer cachexia patients At present, no 2nd-line therapy (or higher) is recommended for pancreatic adenocarcinoma, but often asked for.

Within this clinical trial, we evaluate if parenteral nutrition in combination with chemotherapy in subjects with advanced pancreatic adenocarcinoma have an impact on quality of life?

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histological confirmed advanced pancreatic adenocarcinoma
* At least one previous chemotherapy (gemcitabine-based)
* ≥ 18 years old
* Body weight ≥ 50 and ≤ 95 kg
* BMI ≥ 19
* Negative pregnancy test (females of childbearing potential)
* Willingness to perform double-barrier contraception during study
* Expected life expectancy > 3 months

Exclusion Criteria:

* Major surgery < 4 weeks prior to enrollment
* Weight loss > 2% within the last seven days or caloric intake ≤ 500 kcal expected within the next five days
* PINI-Index > 10
* Pregnancy or breastfeeding
* > 4 weeks of parenteral nutrition within the last 6 months
* Parenteral nutrition < 4 weeks prior to enrollment
* Vulnerable populations (e.g. subjects incapable of giving consent personally)
* Subject selection conflicts with warnings, precautions and contraindications stated for any investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Questionnaire EORTC - Quality of Life | every 1st and 22nd day of a cycle
  The following questionnaires will be given to subjects:
  * EORTC QLQ-C30 (every 1st and 22nd day of a cycle)
  * EORTC QLQ Pan-26 (every 1st and 22nd day of a cycle)

SECONDARY OUTCOMES:
Assessment of nutritional status | every 1st and 22nd day of a cycle)
  * BIA: Phase angle, BCM and Extracellular Mass (ECM)/BCM ratio (every 1st and 22nd day of a cycle)
  * BMI (every 1st and 22nd day of a cycle)
  * Biceps size(every 1st and 22nd day of a cycle)
  * Hand-grip-strength(every 1st and 22nd day of a cycle)
  * PINI-Index (every 1st and 22nd day of a cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Jäger, Prof. Dr., Principal Investigator — University of Heidelberg / National Center for Tumordiseases
Locations (4):
- Germany (4):
  - Onkologische Schwerpunktpraxis und Tagesklinik, Bad Soden
  - Krankenhaus Nordwest Frankfurt, Frankfurt am Main
  - University Hospital of Heidelberg / National Center for Tumordiseases, Heidelberg
  - Asklepios Klinik Weißenfels, Weißenfels

REFERENCES:
- [Background] Marten A, Wente MN, Ose J, Buchler MW, Rotzer I, Decker-Baumann C, Karapanagiotou-Schenkel I, Harig S, Schmidt J, Jager D. An open label randomized multicentre phase IIIb trial comparing parenteral substitution versus best supportive nutritional care in subjects with pancreatic adenocarcinoma receiving 5-FU plus oxaliplatin as 2nd or higher line chemotherapy regarding clinical benefit - PANUSCO. BMC Cancer. 2009 Nov 27;9:412. doi: 10.1186/1471-2407-9-412. PMID 19943918